CLINICAL TRIAL: NCT04253756
Title: A Randomized Trial Examining Plasma Exchange Using the Becton Dickinson (BD) Catheter In an Outpatient Apheresis Unit
Acronym: REPLACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Principal Investigator, Tomas Armendariz, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1363
Record Dates: First submitted 2020-01-25; First posted 2020-02-05 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Plasma Exchange
Keywords: Plasma exchange; Photopheresis; Red blood Cell exchanges

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 18-gauge autogard catheter (No Intervention): Standard of care
- 20-gauge BD Nexiva Diffusics (Experimental): Intervention
  Interventions: Device: 20-gauge BD Nexiva Diffusics

INTERVENTIONS:
Device: 20-gauge BD Nexiva Diffusics — The BD Nexiva Diffusics catheters are suitable for use with power injectors when a direct connection is made.
  Arms: 20-gauge BD Nexiva Diffusics

SUMMARY:
This is a randomized pilot study of therapeutic apheresis procedures (TAP) using the current standard of care catheter (SOC) vs the BD Nexiva Diffusics Catheter. It is a single blinded, randomized study. Data will be used to refine and power a full randomized control trial. For this study, a sample of 33 encounters in each group (total of 66 encounters). The specific aim is to test the hypothesis that the 20-gauge BD Nexiva Diffusics Catheter provides the same efficacy and lower pain level with no increase in adverse events for patients undergoing apheresis treatments.

DETAILED DESCRIPTION:
TAP treats a wide range of disease processes and, in all cases, requires inlet and return venous access to perform the procedure. The goal of TAP is to return the patient to baseline and maintain independence and function. A larger needle (18 gauge) can cause more discomfort to the patient as well as additional scarring. A smaller needle may present less discomfort and scarring to the patient. The goal in the outpatient clinic is to minimize disruption to the patient's routine and help the patient maintain normal activities of daily living.

To accomplish these goals, the outpatient clinic is open Monday thru Friday offering 4 different appointment times. All patients that are referred to the clinic for TAP, first receive a vein evaluation to see if the patient is a candidate for peripheral IV therapy. At the clinic, approximately 68% of the patients TAP's are performed peripherally. This eliminates the risk of a central line infection and any alteration in activities of daily living, such as bathing(Kramer, 2016), (Shang, Ma, Poghosyan, Dowding, & Stone, 2014),(Keller et al., 2018; McDiarmid, 2015).

The hypothesis, is that the 20-gauge BD Nexiva Diffusics catheter provides the same efficacy as current practice with no increase in adverse events for patients undergoing therapeutic apheresis. The results from the study will be significant because if the 20 gauge needle is equally effective for TAP, it can increase the number of patients that would be candidates for peripheral therapy. Therefore, decreasing the need for central venous access, which place the patient at an increased risk of infection. The study is a comparison of 2 types of infusion catheters. The standard of care is an 18-gauge autogard catheter (control group) which will be compared to the 20-gauge BD Nexiva Diffusics (intervention).

P - patients who require therapeutic apheresis procedures (TAP) I - use of 20 guage (20G) BD diffusics catheter during apheresis C - use of 18 G standard of care IV catheter during apheresis O - no difference in efficacy and no increase in safety events

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Speaks and reads English
* A patient of the Apheresis clinic at University of Texas Southwestern University Hospital and Clinics
* Scheduled to receive TAP (therapeutic plasma exchange, red blood cell exchange and extracorporeal Photopheresis) as standard of care

Exclusion Criteria:

* Prisoners
* Persons under the age of 18 years
* Patient who are actively involved in chemotherapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Armendariz, BSN, Principal Investigator — UT Southwestern
Locations (1):
- Zale Lipshy Pavilion, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spires SS, Rebeiro PF, Miller M, Koss K, Wright PW, Talbot TR. Medically Attended Catheter Complications Are Common in Patients With Outpatient Central Venous Catheters. Infect Control Hosp Epidemiol. 2018 Apr;39(4):439-444. doi: 10.1017/ice.2018.8. Epub 2018 Feb 15. PMID 29444733
- [Background] Golestaneh L, Mokrzycki MH. Vascular access in therapeutic apheresis: update 2013. J Clin Apher. 2013 Feb;28(1):64-72. doi: 10.1002/jca.21267. PMID 23420596
- [Background] Kalantari K. The choice of vascular access for therapeutic apheresis. J Clin Apher. 2012;27(3):153-9. doi: 10.1002/jca.21225. Epub 2012 Apr 26. PMID 22535654
- [Background] Keller SC, Williams D, Rock C, Deol S, Trexler P, Cosgrove SE. A new frontier: Central line-associated bloodstream infection surveillance in home infusion therapy. Am J Infect Control. 2018 Dec;46(12):1419-1421. doi: 10.1016/j.ajic.2018.05.016. Epub 2018 Jun 13. No abstract available. PMID 29908838
- [Background] Klimek L, Bergmann KC, Biedermann T, Bousquet J, Hellings P, Jung K, Merk H, Olze H, Schlenter W, Stock P, Ring J, Wagenmann M, Wehrmann W, Mosges R, Pfaar O. Visual analogue scales (VAS): Measuring instruments for the documentation of symptoms and therapy monitoring in cases of allergic rhinitis in everyday health care: Position Paper of the German Society of Allergology (AeDA) and the German Society of Allergy and Clinical Immunology (DGAKI), ENT Section, in collaboration with the working group on Clinical Immunology, Allergology and Environmental Medicine of the German Society of Otorhinolaryngology, Head and Neck Surgery (DGHNOKHC). Allergo J Int. 2017;26(1):16-24. doi: 10.1007/s40629-016-0006-7. Epub 2017 Jan 19. PMID 28217433
- [Background] Shang J, Ma C, Poghosyan L, Dowding D, Stone P. The prevalence of infections and patient risk factors in home health care: a systematic review. Am J Infect Control. 2014 May;42(5):479-84. doi: 10.1016/j.ajic.2013.12.018. Epub 2014 Mar 20. PMID 24656786
- [Background] Putensen D, Leverett D, Patel B, Rivera J. Is peripheral access for apheresis procedures underutilized in clinical practice?-A single centre experience. J Clin Apher. 2017 Dec;32(6):553-559. doi: 10.1002/jca.21508. Epub 2016 Sep 15. PMID 27630072

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: This includes participants where one half was assigned to 18G catheter SOC (control) and the other half be assigned to 20G BD Nexiva Diffusics catheter (intervention). Each participant may participate a maximum of 10 times.
Period: Overall Study
Arm/Group | All Study Participants
Started | 26
Procedure 1: 18 Guage | 12
Procedure 1: 20 Gauge | 14
Procedure 2: 18 Gauge | 9
Procedure 2: 20 Gauge | 7
Procedure 3: 18 Gauge | 6
Procedure 3: 20 Gauge | 5
Procedure 4: 18 Gauge | 5
Procedure 4: 20 Gauge | 3
Procedure 5: 18 Gauge | 2
Procedure 5: 20 Gauge | 3
Procedure 6: 18 Gauge | 1
Procedure 6: 20 Gauge | 2
Procedure 7: 18 Gauge | 1
Procedure 7: 20 Gauge | 1
Procedure 8: 18 Gauge | 0
Procedure 8: 20 Gauge | 2
Completed | 21
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Due to the cross over study design, participants are represented as one Baseline group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Assigned Intervention as Measured by Plasma Hemoglobin Value
Description: Efficacy of assigned intervention is measured by comparing the mean plasma hemoglobin values by group. Plasma hemoglobin test will be run on each patient to test for hemolysis (destruction of red blood cells which leads to the release of hemoglobin from the red blood cells into the blood plasma) which will be scored dichotomously as present or absent.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- 18G Catheter SOC (Control): The standard of care is an 18-gauge autogard catheter (control group)
- 20-gauge BD Nexiva Diffusics (Intervention): 20-gauge BD Nexiva Diffusics: The BD Nexiva Diffusics catheters are suitable for use with power injectors when a direct connection is made.
Arm/Group | 18G Catheter SOC (Control) | 20-gauge BD Nexiva Diffusics (Intervention)
Number analyzed (Participants) | 13 | 13
g/dL | 16.8 (9.64) | 17.3 (12.4)
Statistical Analysis 1: Comparison: 18G Catheter SOC (Control) vs 20-gauge BD Nexiva Diffusics (Intervention); Test type: Non-Inferiority — The margin of non-inferiority (Delta) was 5g/dl; p = 0.87, ANOVA; Mean Difference (Final Values) = 0.5

2. Primary Outcome: Efficacy of Assigned Intervention as Measured by the Amount of Time (Minutes) Required to Complete a TAP
Description: Efficacy of assigned intervention is measured by comparing the time to complete the TAP in minutes and comparing the two treatment groups.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 18G Catheter SOC (Control) | 20-gauge BD Nexiva Diffusics (Intervention)
Number analyzed (Participants) | 13 | 13
minutes | 90.1 (14.3) | 86.9 (13.2)
Statistical Analysis 1: Comparison: 18G Catheter SOC (Control) vs 20-gauge BD Nexiva Diffusics (Intervention); Test type: Non-Inferiority — The non-inferiority margin (Delta) was 10 minutes of run time, no other key parameters; p = 0.32, ANOVA; Mean Difference (Final Values) = 3.2

3. Primary Outcome: Number of Adverse Events Experienced by Participants in Each Group
Description: Number of adverse events experienced by participants in each group is being compared here.
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | 18G Catheter SOC (Control) | 20-gauge BD Nexiva Diffusics (Intervention)
Number analyzed (Participants) | 13 | 13
events | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing a Return Pressure >400 mmHg
Description: Number of participants experiencing a return pressure >400 mmHg when the return catheter occupies <45% of the inner-lumen diameter is being measured. The suggested standard is that a catheter occupies < 45% of the inner-lumen diameter (measured with ultrasound). Return pressures >400 mm Hg are considered problematic.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | 18G Catheter SOC (Control) | 20-gauge BD Nexiva Diffusics (Intervention)
Number analyzed (Participants) | 13 | 13
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: When the return rate is out of the SOC parameters the SOC apheresis equipment (Optia or Cellex) will alarm. If the alarm sounds 3 times the RN will decrease inlet rate by 5 ml/sec until the minimum threshold is reached (if needed), which is 50 ml/sec for plasma exchange and 35 ml/sec for RBC exchange and 20 ml/sec for photopheresis. If the alarm continues to when the minimum threshold is reached the catheter will be replaced with the SOC 18-gauge catheter.
Arm/Group | 18-gauge Autogard Catheter | 20-gauge BD Nexiva Diffusics
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04253756/Prot_SAP_001.pdf